CLINICAL TRIAL: NCT00196235
Title: Innovative Stratification of Arrhythmic Risk (ISAR-Trial): Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Other Study IDs: GE IDE No. R00295
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2005-09

CONDITIONS: Myocardial Infarction
Keywords: Assessment, Risk; Diabetes mellitus; Autonomic nervous system
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study was to evaluate the performance of established and new risk predictors in predicting mortality in post-infarction patients suffering from diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

acute myocardial infarction, presence of sinusrhythm

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmidt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Petra Barthel, MD, Study Director — Deutsches Herzzentrum Muenchen; Axel Bauer, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Schmidt G, Malik M, Barthel P, Schneider R, Ulm K, Rolnitzky L, Camm AJ, Bigger JT Jr, Schomig A. Heart-rate turbulence after ventricular premature beats as a predictor of mortality after acute myocardial infarction. Lancet. 1999 Apr 24;353(9162):1390-6. doi: 10.1016/S0140-6736(98)08428-1. PMID 10227219
- [Result] Barthel P, Schneider R, Bauer A, Ulm K, Schmitt C, Schomig A, Schmidt G. Risk stratification after acute myocardial infarction by heart rate turbulence. Circulation. 2003 Sep 9;108(10):1221-6. doi: 10.1161/01.CIR.0000088783.34082.89. Epub 2003 Aug 25. PMID 12939209
- [Result] Makikallio TH, Barthel P, Schneider R, Bauer A, Tapanainen JM, Tulppo MP, Schmidt G, Huikuri HV. Prediction of sudden cardiac death after acute myocardial infarction: role of Holter monitoring in the modern treatment era. Eur Heart J. 2005 Apr;26(8):762-9. doi: 10.1093/eurheartj/ehi188. Epub 2005 Mar 18. PMID 15778204
- [Result] Bauer A, Guzik P, Barthel P, Schneider R, Ulm K, Watanabe MA, Schmidt G. Reduced prognostic power of ventricular late potentials in post-infarction patients of the reperfusion era. Eur Heart J. 2005 Apr;26(8):755-61. doi: 10.1093/eurheartj/ehi101. Epub 2005 Jan 26. PMID 15673543